CLINICAL TRIAL: NCT00982592
Title: A Randomized, Double Blind Placebo Controlled Phase 2 Study of FOLFOX Plus or Minus GDC-0449 in Patients With Advanced Gastric and Gastroesophageal Junction (GEJ) Carcinoma
Brief Title: Combination Chemotherapy With or Without Vismodegib in Treating Patients With Advanced Stomach Cancer or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2011-01425; NCI-2011-01425 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 09-0356; CDR0000655339; NYU 09-0356 (Other: New York University Langone Medical Center); 8376 (Other: CTEP); N01CM00038 (NIH); N01CM00071 (NIH); P30CA016087 (NIH); N01CM00070 (NIH)
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-08

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Adenocarcinoma of the Stomach; Recurrent Gastric Cancer; Stage IIIA Gastric Cancer; Stage IIIB Gastric Cancer; Stage IIIC Gastric Cancer; Stage IV Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Leucovorin; Fluorouracil; HhAntag691

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (FOLFOX regimen and placebo) (Experimental): Patients receive FOLFOX chemotherapy comprising oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil bolus and then IV over 46-48 hours on day 1. Patients also receive placebo PO QD on days 1-14. Courses repeat every 2 weeks in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: oxaliplatin; Drug: leucovorin calcium; Drug: fluorouracil; Other: placebo; Other: laboratory biomarker analysis
- Arm II (FOLFOX regimen and vismodegib) (Experimental): Patients receive FOLFOX chemotherapy as in arm I. Patients also receive vismodegib PO on days 1-14. Courses repeat every 2 weeks in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: oxaliplatin; Drug: leucovorin calcium; Drug: fluorouracil; Drug: vismodegib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm I (FOLFOX regimen and placebo)
Drug: vismodegib — Given PO
  Other Names: Erivedge; GDC-0449; Hedgehog antagonist GDC-0449
  Arms: Arm II (FOLFOX regimen and vismodegib)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies combination chemotherapy when given together with vismodegib to see how well it works compared with combination chemotherapy without vismodegib in treating patients with advanced stomach cancer or gastroesophageal junction cancer. Drugs used in chemotherapy, such as oxaliplatin, leucovorin calcium, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Vismodegib may stop the growth of stomach or gastroesophageal junction cancer by blocking the growth of new blood vessels necessary for tumor growth. It is not yet known whether combination chemotherapy is more effective when given with or without vismodegib in treating stomach cancer and gastroesophageal junction cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the addition of GDC-0449 (vismodegib) to FOLFOX (fluorouracil, leucovorin calcium, oxaliplatin) chemotherapy improves median progression free survival (PFS) in the first line treatment of patients with advanced gastric and gastroesophageal junction (GEJ) adenocarcinoma.

SECONDARY OBJECTIVES:

I. To determine if the addition of GDC-0449 to FOLFOX chemotherapy affects overall survival.

II. To determine if the addition of GDC-0449 to FOLFOX chemotherapy affects response rate.

III. To determine if the addition of GDC-0449 to FOLFOX chemotherapy affects toxicity rates in the first line treatment of patients with advanced gastric and GEJ adenocarcinoma.

TERTIARY OBJECTIVES:

I. To determine the level of baseline hedgehog pathway activation and correlate with clinical outcome and response to treatment with GDC-0449.

II. In those patients who consent to repeat biopsy at week 4-5, hedgehog pathway expression will again be assessed (every attempt will be made to obtain repeat biopsy from the same site as the initial biopsy) and compared to baseline values and clinical outcome.

III. To determine a primary gastric cancer gene expression profile that may predict response to GDC-0449.

IV. To determine if serum shed collagen epitopes correlate with clinical outcome and may be used to assess efficacy of GDC-0449 treatment.

V. To determine if circulating endothelial progenitor cells (EPC)'s correlate with treatment response and may be used to assess efficacy of GDC-0449 treatment.

VI. To determine if hedgehog pathway expression is downregulated in EPC's following treatment with GDC-0449.

VII. To determine if serum expression of vascular endothelial growth factor (VEGF), transforming growth factor (TGF)-beta, and insulin-like growth factor binding protein (IGFBP) 3 correlate with clinical outcome and may be used to assess efficacy of GDC-0449 treatment.

VIII. To determine if human epidermal growth factor receptor 2 (Her2) expression is predictive in assessing the efficacy of GDC-0449 treatment. Of note, Her2 status will be collected retrospectively for those patients who were tested as part of standard of care established in October 2010.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive FOLFOX chemotherapy comprising oxaliplatin intravenously (IV) over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV over 46-48 hours on day 1. Patients also receive placebo orally (PO) once daily (QD) on days 1-14.

ARM II: Patients receive FOLFOX chemotherapy as in Arm I. Patients also receive vismodegib PO on days 1-14. In both arms, treatment repeats every 2 weeks in the absence of unacceptable toxicity or disease progression.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed gastric or gastroesophageal junction (GEJ) adenocarcinoma not amenable to surgical resection
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan
* No prior chemotherapy for advanced disease; patients may have receive adjuvant chemotherapy or chemoradiation if > 6 months has elapsed since completion of treatment
* Life expectancy of greater than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status < 2 (Karnofsky > 70%)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal (=< 5.0 X institutional upper limit of normal with presence of liver metastases)
* Creatinine =< 1.5 X institutional upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Baseline imaging studies performed =< 28 days of study registration; the treating investigator will determine the appropriate imaging studies, which may include CT scan, magnetic resonance imaging (MRI), and/or fludeoxyglucose F 18 (FDG)-positron emission tomography (PET)/CT
* Must be willing to provide blood and tissue samples for research purposes; patient has the right to later withdraw consent for research studies and/or tissue specimens
* Patients must agree to placement of a central venous catheter for chemotherapy administration
* Patients must be able to swallow whole capsules
* Patients taking medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin), must be on a stable, therapeutic dose and have close monitoring of their levels
* Women of child-bearing potential and men must use two forms of contraception (i.e., barrier contraception and one other method of contraception) at least 4 weeks prior to study entry, for the duration of study participation, and for at least 12 months post-treatment; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Pregnancy testing: women of childbearing potential are required to have a negative serum pregnancy test (with a sensitivity of at least 25 mIU/mL) within 10-14 days and within 24 hours prior to the first dose of GDC-0449/placebo (serum or urine); a pregnancy test (serum or urine) will be administered every 4 weeks if their menstrual cycles are regular or every 2 weeks if their cycles are irregular while on study within the 24-hour period prior to the administration of GDC-0449/placebo; a positive urine test must be confirmed by a serum pregnancy test; prior to dispensing GDC-0449/placebo, the investigator must confirm and document the patient's use of two contraceptive methods, dates of negative pregnancy test, and confirm the patient's understanding of the teratogenic potential of GDC-0449/placebo
* Female subjects of childbearing potential are defined as follows:

  * Patients with regular menses
  * Patients, after menarche with amenorrhea, irregular cycles, or using a contraceptive method that precludes withdrawal bleeding
  * Women who have had tubal ligation
* Female subjects may be considered to NOT be of childbearing potential for the following reasons:

  * The patient has undergone hysterectomy and/or bilateral oophorectomy.
  * The patient is post-menopausal defined by amenorrhea for at least 1 year in a woman > 45 years old
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 6 months prior to entering the study
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to GDC-0449, 5-fluorouracil or oxaliplatin
* GDC-0449 inhibits cytochrome P450, family 2, subfamily C, polypeptide 8 (CYP2C8), cytochrome P450, family 2, subfamily C, polypeptide 9 (CYP2C9), and cytochrome P450, family 2, subfamily C, polypeptide 19 (CYP2C19) drug metabolism enzymes in vitro at concentrations that may be clinically relevant; therefore, caution should be exercised when dosing GDC-0449 concurrently with medications that are substrates of CYP2C8, CYP2C9, and CYP2C19 and have narrow therapeutic windows
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption
* Patients unable to swallow whole capsules
* Patients with clinically active liver disease, including viral or other hepatitis or cirrhosis are ineligible
* Patients with uncontrolled hypocalcemia, hypomagnesemia, hyponatremia or hypokalemia defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation are excluded from this study
* Pre-existing > grade 1 peripheral sensory neuropathy
* Previous or concurrent malignancy; exceptions: treated basal cell or squamous cell skin cancer, in situ cervical cancer, or lobular carcinoma in situ in one breast; or other cancer which the patient has been disease-free ≥5 years
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with GDC-0449
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2009-09; Primary Completion 2012-04 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Cohen, Principal Investigator — NYU Langone Health
Locations (30):
- United States (30):
  - University of California at Davis Cancer Center, Sacramento, California
  - University of Chicago, Chicago, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University Medical Center, Indianapolis, Indiana
  - University of Michigan University Hospital, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Beth Israel Medical Center, New York, New York
  - New York University Langone Medical Center, New York, New York
  - Saint Luke's Roosevelt Hospital Center - Saint Luke's Division, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - New York Cancer Consortium, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Virginia Commonwealth University, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From October 2009 to February 2012, 124 patients were enrolled from multi sites to this study.
Period: Overall Study
Arm/Group | Arm I (FOLFOX Regimen and Placebo) | Arm II (FOLFOX Regimen and Vismodegib)
Started | 64 | 60
Treatment Received | 63 | 52
Completed | 33 (patients who were off treatment due to disease progression) | 27 (patients who were off treatment due to disease progression)
Not Completed | 31 | 33

BASELINE CHARACTERISTICS:
Population: all the patients enrolled to the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (FOLFOX Regimen and Placebo) | Arm II (FOLFOX Regimen and Vismodegib) | Total
Number analyzed (Participants) | 64 | 60 | 124
Age, Continuous [Median (Full Range); unit: years] | 61.5 [25 to 77] | 57.5 [29 to 74] | 60 [25 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 21 | 32
  Male | 53 | 39 | 92
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 50 | 42 | 92
  Asian | 3 | 6 | 9
  African American | 6 | 4 | 10
  Hispanic | 4 | 8 | 12
  Nor reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 64 | 60 | 124

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-free Survival (PFS)
Description: PFS is defined as the time from randomization until objective tumor progression or death from any cause and is evaluated per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Time Frame: up to 4 years
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (FOLFOX Regimen and Placebo) | Arm II (FOLFOX Regimen and Vismodegib)
Number analyzed (Participants) | 64 | 60
months | 8.77 [5.65 to 10.61] | 8.35 [5.55 to 10.61]
Statistical Analysis 1: Comparison: Arm I (FOLFOX Regimen and Placebo) vs Arm II (FOLFOX Regimen and Vismodegib); Test type: Superiority or Other; p = 0.874, Log Rank; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.70 to 1.54]

2. Secondary Outcome: Objective Response Rate
Description: Defined as the percentage of the patients who had complete response (CR) or partial response (PR) per RECIST 1.1.
Time Frame: Up to 4 years
Population: Intent-to-treat population
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (FOLFOX Regimen and Placebo) | Arm II (FOLFOX Regimen and Vismodegib)
Number analyzed (Participants) | 64 | 60
percentage of patients | 44 | 37

3. Secondary Outcome: Overall Survival
Description: Defined as time from randomization day until death from any cause.
Time Frame: up to 4 years
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (FOLFOX Regimen and Placebo) | Arm II (FOLFOX Regimen and Vismodegib)
Number analyzed (Participants) | 64 | 60
months | 15.38 [12.32 to 19.52] | 12.12 [10.28 to 17.77]
Statistical Analysis 1: Comparison: Arm I (FOLFOX Regimen and Placebo) vs Arm II (FOLFOX Regimen and Vismodegib); Test type: Superiority or Other; p = 0.253, Log Rank; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [0.83 to 2.05]

4. Secondary Outcome: Incidence of Toxicities (Grade 3 and Higher)
Description: Defined as percentage of patients who experienced a toxicity with grade 3 or higher related to the protocol therapy. Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0
Time Frame: Up to 4 years
Population: All the patients who started the treatment.
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (FOLFOX Regimen and Placebo) | Arm II (FOLFOX Regimen and Vismodegib)
Number analyzed (Participants) | 63 | 52
percentage of patients
  Neuropathy (sensory) | 13 | 19
  Fatigue | 10 | 15
  Thrombosis | 11 | 14
  Nausea | 8 | 8
  Hemorrhage_GI | 11 | 8
  Vomiting | 6 | 8
  Dehydration | 6 | 8
  Neutropenia | 32 | 50
  Febrile neutropenia | 5 | 2
  Anemia | 10 | 10
  Thrombocytopenia | 0 | 6
  Hypokalemia | 5 | 10
  Hyperglycemia | 10 | 4
  Hyponatremia | 10 | 2

5. Secondary Outcome: Incidence of Toxicities (grades1 and 2)
Description: Defined as percentage of patients who experienced a toxicity with grade 1 or 2 (worst grade) related to the protocol therapy. Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0.
Time Frame: Up to 4 years
Population: All the patients who started the treatment.
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (FOLFOX Regimen and Placebo) | Arm II (FOLFOX Regimen and Vismodegib)
Number analyzed (Participants) | 63 | 52
percentage of patients
  Neuropathy (sensory) | 56 | 62
  Fatigue | 54 | 73
  Diarrhea | 48 | 40
  Nausea | 54 | 71
  Dysguesia | 16 | 42
  Vomiting | 38 | 37
  Anorexia | 41 | 35
  Weight loss | 30 | 29
  Leukocytes | 57 | 46
  Anemia | 51 | 60
  Thrombocytopenia | 57 | 56
  Hypoalbuminemia | 52 | 40
  Hyperglycemia | 41 | 37
  Elevated AST | 29 | 46

ADVERSE EVENTS:
Time Frame: Up to 4 years.
Description: All the adverse events above the reporting threshold are reported here regardless of attributions. Sixty three patients on the placebo arm and 52 on the Vismodegib arm started treatments; 1 and 8 patients did not receive treatments, respectively.
Arm/Group | Arm I (FOLFOX Regimen and Placebo) | Arm II (FOLFOX Regimen and Vismodegib)
Serious Adverse Events (participants affected / at risk) | 24/63 | 20/52
Other Adverse Events (participants affected / at risk) | 63/63 | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (FOLFOX Regimen and Placebo) (N=63) | Arm II (FOLFOX Regimen and Vismodegib) (N=52)
Ascites (non-malignant) (Gastrointestinal disorders) | 1 | 0
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 | 1
Cardiac General - Other (Specify, __)SINUS BRADYCARDIA (Cardiac disorders) | 0 | 1
Cardiac ischemia/infarction (Cardiac disorders) | 1 | 0
CNS cerebrovascular ischemia (Nervous system disorders) | 0 | 1
Death not associated with CTCAE term: Death NOS (General disorders) | 3 | 2
Death not associated with CTCAE term: Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Dehydration (Gastrointestinal disorders) | 3 | 3
Diarrhea (Gastrointestinal disorders) | 3 | 1
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 | 0
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 | 3
Febrile neutropenia (Infections and infestations) | 2 | 1
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 | 3
Gastrointestinal - Other (Specify, __)MALIGNANT ASCITES (Gastrointestinal disorders) | 0 | 1
Gastrointestinal - Other (Specify, __)GASTRIC PERFORATION (Gastrointestinal disorders) | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 1 | 0
Hemorrhage, GI: Esophagus (Gastrointestinal disorders) | 1 | 0
Hemorrhage, GI: Stomach (Gastrointestinal disorders) | 1 | 2
Hemorrhage, GI: Lower GI NOS (Gastrointestinal disorders) | 1 | 0
Hemorrhage, GI: Upper GI NOS (General disorders) | 3 | 0
Hepatobiliary/Pancreas - Other (Specify, __)VENO-OCCLUSIVE DISEASE (Hepatobiliary disorders) | 1 | 0
Hypotension (Cardiac disorders) | 1 | 0
Infection - Other (Specify, __)PLEURAL ABSCESS (Infections and infestations) | 1 | 0
Infection - Other (Specify, __)THRUSH (Infections and infestations) | 1 | 0
Infection with Grade 3 or 4 neutrophils: Lung (pneumonia) (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Catheter-related (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Kidney (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Lung (pneumonia) (Infections and infestations) | 2 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Wound (Infections and infestations) | 1 | 0
Infection with unknown ANC: Lung (pneumonia) (Infections and infestations) | 1 | 0
Infection with unknown ANC: Pleura (empyema) (Infections and infestations) | 1 | 0
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Mental status (Nervous system disorders) | 0 | 1
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-lower (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-upper (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal/Soft Tissue - Other (Specify, __)KNEE PAIN AND SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3
Neurology - Other (Specify, __)DECREASED RESPONSIVENESS AFTER SEDATION (Nervous system disorders) | 1 | 0
Neuropathy: sensory (Nervous system disorders) | 1 | 0
Neuropathy: motor (Nervous system disorders) | 0 | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 | 4
Obstruction, GU: Ureter (Renal and urinary disorders) | 0 | 1
Obstruction, GI: Colon (Gastrointestinal disorders) | 1 | 0
Pain: Abdomen NOS (Gastrointestinal disorders) | 1 | 3
Pain: Chest wall (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain: Intestine (Gastrointestinal disorders) | 1 | 0
Pain: Joint (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain: Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Portal vein flow (Vascular disorders) | 1 | 0
Pulmonary/Upper Respiratory - Other (Specify, __)MALIGNANT PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Stricture/stenosis (including anastomotic), GI: Stomach (Gastrointestinal disorders) | 0 | 1
Syncope (fainting) (Nervous system disorders) | 1 | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 5 | 2
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (FOLFOX Regimen and Placebo) (N=63) | Arm II (FOLFOX Regimen and Vismodegib) (N=52)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 35 | 21
Alkaline phosphatase (Metabolism and nutrition disorders) | 22 | 22
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 4 | 2
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 0 | 5
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 11 | 23
Anorexia (Gastrointestinal disorders) | 27 | 20
Ascites (non-malignant) (Gastrointestinal disorders) | 3 | 0
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 20 | 23
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 2 | 7
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 8 | 4
Blood/Bone Marrow - Other (Specify, __)LOW EOSINOPHILS (Blood and lymphatic system disorders) | 3 | 0
Blood/Bone Marrow - Other (Specify, __)HIGH LYMPHOCYTES (Blood and lymphatic system disorders) | 3 | 0
Blood/Bone Marrow - Other (Specify, __)LOW EOSINOPHILS (Blood and lymphatic system disorders) | 2 | 0
Blood/Bone Marrow - Other (Specify, __)MONOCYTOSIS (Blood and lymphatic system disorders) | 4 | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 19 | 9
Cheilitis (Skin and subcutaneous tissue disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 24 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 9
Creatinine (Metabolism and nutrition disorders) | 3 | 4
Dehydration (Gastrointestinal disorders) | 4 | 6
Diarrhea (Gastrointestinal disorders) | 32 | 21
Distension/bloating, abdominal (Gastrointestinal disorders) | 0 | 5
Dizziness (Nervous system disorders) | 13 | 12
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 3 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 3
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 11 | 12
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 13 | 8
Edema:limb (Blood and lymphatic system disorders) | 9 | 4
Fatigue (asthenia, lethargy, malaise) (General disorders) | 44 | 44
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 7 | 5
Fracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Flatulence (Gastrointestinal disorders) | 2 | 0
Flu-like syndrome (General disorders) | 3 | 0
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 2 | 2
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 31 | 22
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 3 | 5
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 7 | 9
Heartburn/dyspepsia (Gastrointestinal disorders) | 4 | 10
Hemoglobin (Blood and lymphatic system disorders) | 37 | 34
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Blood and lymphatic system disorders) | 3 | 2
Hemorrhage, GI: Esophagus (Gastrointestinal disorders) | 0 | 2
Hemorrhage, GI: Rectum (Gastrointestinal disorders) | 2 | 0
Hemorrhage, pulmonary/upper respiratory: Nose (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypertension (Cardiac disorders) | 4 | 0
Hypotension (Cardiac disorders) | 3 | 0
Infection - Other (Specify, __)THRUSH (Infections and infestations) | 4 | 3
Infection with normal ANC or Grade 1 or 2 neutrophils: External ear (otitis externa) (Infections and infestations) | 2 | 0
Infection with unknown ANC: Urinary tract NOS (Infections and infestations) | 0 | 2
INR (International Normalized Ratio of prothrombin time) (Investigations) | 0 | 2
Insomnia (General disorders) | 5 | 11
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 40 | 29
Lymphopenia (Blood and lymphatic system disorders) | 23 | 16
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 | 4
Memory impairment (Nervous system disorders) | 2 | 0
Metabolic/Laboratory - Other (Specify, __)LOW CO2 (Metabolism and nutrition disorders) | 2 | 0
Metabolic/Laboratory - Other (Specify, __)TOTAL PROTEIN DECREASED (Metabolism and nutrition disorders) | 4 | 0
Mood alteration: Anxiety (Nervous system disorders) | 4 | 3
Mood alteration: Depression (Nervous system disorders) | 4 | 6
Mucositis/stomatitis (clinical exam): Oral cavity (Gastrointestinal disorders) | 12 | 7
Mucositis/stomatitis (functional/symptomatic): Oral cavity (Gastrointestinal disorders) | 9 | 4
Muscle weakness, generalized or specific area (not due to neuropathy): Whole body/generalized (Musculoskeletal and connective tissue disorders) | 3 | 0
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 40 | 41
Neurology - Other (Specify, __)COLD SENSITIVITY (Nervous system disorders) | 5 | 4
Neuropathy: motor (Nervous system disorders) | 4 | 3
Neuropathy: sensory (Nervous system disorders) | 42 | 42
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 28 | 33
Pain - Other (Specify, __)GROIN (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain - Other (Specify, __)RIB (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain: Abdomen NOS (Gastrointestinal disorders) | 23 | 4
Pain: Back (Musculoskeletal and connective tissue disorders) | 9 | 4
Pain: Bone (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain: Chest wall (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain: Chest/thorax NOS (General disorders) | 6 | 4
Pain: Esophagus (Gastrointestinal disorders) | 2 | 0
Pain: Extremity-limb (Musculoskeletal and connective tissue disorders) | 9 | 7
Pain: Head/headache (Nervous system disorders) | 6 | 8
Pain: Joint (Musculoskeletal and connective tissue disorders) | 6 | 6
Pain: Muscle (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain: Neck (Musculoskeletal and connective tissue disorders) | 2 | 5
Pain: Oral cavity (Gastrointestinal disorders) | 6 | 2
Pain: Stomach (Gastrointestinal disorders) | 3 | 2
Pain: Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Palpitations (Cardiac disorders) | 3 | 0
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 5 | 3
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 2
Platelets (Blood and lymphatic system disorders) | 36 | 32
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 6 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 22 | 12
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 | 2
Pulmonary/Upper Respiratory - Other (Specify, __)RUNNY NOSE (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6 | 6
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2 | 2
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 3 | 4
Rigors/chills (General disorders) | 3 | 6
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 2 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 22 | 17
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 10 | 24
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 6
Tremor (Nervous system disorders) | 0 | 2
Urinary frequency/urgency (Renal and urinary disorders) | 3 | 3
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 3 | 0
Vision-blurred vision (Eye disorders) | 5 | 2
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 28 | 22
Weight loss (General disorders) | 19 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less